CLINICAL TRIAL: NCT05361369
Title: A Single Center, Single Arm, Single Dose, Bioavailability Study of EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule (a Fixed Dose Combination of 600 mg Fenticonazole Nitrate + 1000 mg Tinidazole + 100 mg Lidocaine) in 18 Healthy Female Subjects
Brief Title: Bioavailability Study of EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exeltis Turkey (Industry)
Collaborators: Monitor CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MON837.130.6
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Bioavailability
Keywords: fenticonazole nitrate; tinidazole; lidocaine; fixed-dose combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule (Experimental): Fixed dose combination of 600 mg fenticonazole nitrate + 1000 mg tinidazole + 100 mg lidocaine vaginal ovule will be administered once as a single dose during a single-period.
  Interventions: Drug: EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule

INTERVENTIONS:
Drug: EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule — Fixed dose combination of 600 mg fenticonazole nitrate + 1000 mg tinidazole + 100 mg lidocaine

SUMMARY:
A single dose of the study drug will be administered to healthy female subjects in a single period to obtain pharmacokinetic parameters for each active ingredient.

DETAILED DESCRIPTION:
The study drug, EVEGYN 600 mg/1000 mg/100 mg Vaginal Ovule, is a fixed-dose combination of 600 mg fenticonazole nitrate + 1000 mg tinidazole + 100 mg lidocaine. It is manufactured by Exeltis İlaç San. ve Tic. A.Ş., Turkey. It is an antibacterial and antifungal medication that will be used in the treatment of common vaginitis (e.g. bacterial vaginosis, candidal vulvovaginitis). Its efficacy and safety were previously evaluated in a Phase III clinical trial. In this single-center, single-arm, single-dose, bioavailability study, pharmacokinetic parameters for each active ingredient will be evaluated in 18 healthy female subjects following intravaginal administration of this fixed-dose combination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female adult subject with age of ≥ 18 and ≤ 55 years who have a regular menstrual cycle (at least 10 times a year),
* Subject with a body weight ≥ 50 kg and body mass index between 16 and 30 kg/m2
* Informed consent signed by the subject.

Exclusion Criteria:

* Positive rapid antigen or polymerase chain reaction test result for COVID-19
* Pregnancy and/or breastfeeding, or subject who doesn't accept not to get pregnant during the study
* Known hypersensitivity to active ingredients (including their derivatives) of the study medication
* Postmenopausal women

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
AUC0-72 | 0-72 hours
  Area under the plasma concentration-time profile from time zero to 72 hours post dose based on observed plasma concentrations for each analyte
Cmax | 0-72 hours
  Maximum observed plasma concentration for each analyte

SECONDARY OUTCOMES:
Tmax | 0-72 hours
  Time to reach maximum plasma concentration for each analyte
AUC0-inf | 0-72 hours
  Area under the plasma concentration-time profile from time zero to infinity based on observed plasma concentrations for each analyte
T1/2 | 0-72 hours
  Half-life for each analyte
Lambda-z | 0-72 hours
  Elimination rate constant for each analyte

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hakan Çetinsaya İyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP), Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No